CLINICAL TRIAL: NCT03545282
Title: ALMA: A Randomized Control Trial of an Intervention to Reduce Mental Health Disparities in Mexican Immigrant Women
Brief Title: Intervention Trial to Reduce Mental Health Disparities in Latina Immigrant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, India Ornelas, Associate Professor, School of Public Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00003331; R01MD012230 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-06-04 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Stress; Depression; Anxiety
Keywords: Mental Health; Minority Health; Latina
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and outcomes assessor will not have knowledge of the interventions assigned to individual participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALMA Intervention Group (Experimental): Amigas Latinas Motivando el Alma (ALMA). This group receives the intervention after baseline assessment.
  Interventions: Behavioral: Amigas Latinas Motivando el Alma (ALMA)
- ALMA Delayed Intervention Control Group (Other): Amigas Latinas Motivando el Alma (ALMA). This group receives the intervention five months after the baseline assessment (after the post-intervention, and 3 month assessments have been completed).
  Interventions: Behavioral: Amigas Latinas Motivando el Alma (ALMA)

INTERVENTIONS:
Behavioral: Amigas Latinas Motivando el Alma (ALMA) — In a series of 8 weekly sessions, the program uses a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. Over the course of the eight ALMA sessions, 25 women are (1) engaged in activities to identify coping strategies they are currently using and encouraged to continue to use them; (2) introduced to new coping strategies (e.g. mindfulness techniques, increased social ties and social support); and, (3) provided resources for seeking additional help if needed.
  Due to COVID-19 pandemic, the intervention was changed to online synchronous delivery via Zoom over 6 weekly sessions.

SUMMARY:
Latina immigrant women are particularly vulnerable to depression and anxiety due to the social and economic stressors they face, including high levels of poverty, low levels of education, family obligations, exposure to violence, and limited access to community resources. ALMA aims to prevent and reduce depression and anxiety among Latina immigrant women. Women attend 8 weekly sessions in a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. The intervention aims to increase participants' social ties and the social support they receive from other Latina immigrant women. The program also helps decrease the stigma associated with mental health and connects women to mental health services when needed.

DETAILED DESCRIPTION:
The proposed study aims to test the efficacy of the Amigas Latinas Motivando el Alma (ALMA) intervention in a randomized control trial. ALMA is an 8-week program offered in a group format to teach women new coping strategies and enhance their social ties and social support to prevent and reduce their depression and anxiety. Aim 1 of the proposed study is to refine the ALMA intervention and study procedures, using information learned from focus groups and cognitive interviews with Mexican immigrant women. Aim 2 is to determine the efficacy of the ALMA intervention to reduce depressive and anxiety symptoms using a randomized control study design. We will recruit women from community-based organizations serving Latino immigrants to participate in the program, which will be offered in community settings. We will assess process outcomes of recruitment, retention, fidelity, and participant satisfaction through observations and in-depth interviews with participants. We will assess the efficacy of the intervention by comparing changes in women's depressive and anxiety symptoms in the intervention and attention control groups at four time points (pre-intervention, post-intervention, 6 months, 9 months). Aim 3 is to assess the potential impact of the intervention on both individual (stigma, stress, coping strategies) and interpersonal (social support, social ties) factors, and whether the impact of the intervention is mediated by these factors. The research team includes investigators in psychology, medicine, social work and public health, as well as community-based organizations serving Latina immigrants. The study uses rigorous methods to test an innovative program that integrates both culturally relevant and evidenced-based strategies to address significant mental health disparities in a high-risk and underserved population. Findings will help inform future research and practice. Given the growth of the Latino population, identifying interventions that reduce mental health disparities among Mexican immigrant women can have a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for study participation, participants must be at least 18 years of age, female, speak Spanish, must self-identify as Latina, and have been born outside of the United States.

Exclusion Criteria:

* Participant screened for high levels of depressive symptoms (as indicated by a score of 20 or higher on the PHQ-9) which indicates severe symptoms. Participants with scores above 20 were referred to the licensed mental health counselor on the study team. If these women are not already receiving mental health treatment, they will be referred to mental health providers offering low-cost services in Spanish. The counselor will discuss participation in the program with the potential participants and make the final determination about their ability to participate based on the care they are currently receiving and the severity of their symptoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men will not be included in the study. Participation is limited to this population because the research question addressed is relevant only to Latina women and the mental health concerns of this community.
Enrollment: 226 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: India J Ornelas, PhD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Casa Latina, Seattle, Washington
  - El Centro de la Raza, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abarca GJ, Tornberg-Belanger SN, Ryan D, Price C, Rao D, Ornelas IJ. Understanding the Relationship Between Social Stressors, Trauma, and Somatic Symptoms Among Latina Immigrant Women. J Racial Ethn Health Disparities. 2023 Feb;10(1):387-394. doi: 10.1007/s40615-022-01230-9. Epub 2022 Mar 7. PMID 35257311
- [Background] Ornelas IJ, Tornberg-Belanger S, Balkus JE, Bravo P, Perez Solorio SA, Perez GE, Tran AN. Coping With COVID-19: The Impact of the Pandemic on Latina Immigrant Women's Mental Health and Well-being. Health Educ Behav. 2021 Dec;48(6):733-738. doi: 10.1177/10901981211050638. Epub 2021 Oct 21. PMID 34672827
- [Background] Ryan D, Tornberg-Belanger SN, Perez G, Maurer S, Price C, Rao D, Chan KCG, Ornelas IJ. Stress, social support and their relationship to depression and anxiety among Latina immigrant women. J Psychosom Res. 2021 Oct;149:110588. doi: 10.1016/j.jpsychores.2021.110588. Epub 2021 Jul 30. PMID 34371256
- [Result] Ornelas IJ, Rao D, Price C, Chan G, Tran A, Aisenberg G, Perez G, Maurer S, Nelson AK. Promoting mental health in Latina immigrant women: Results from the Amigas Latinas Motivando el Alma intervention trial. Soc Sci Med. 2023 Mar;321:115776. doi: 10.1016/j.socscimed.2023.115776. Epub 2023 Feb 16. PMID 36809698
- [Result] Ornelas IJ, Perez G, Maurer S, Gonzalez S, Childs V, Price C, Nelson AK, Perez Solorio SA, Tran A, Rao D. Amigas Latinas Motivando el Alma: In-Person and Online Delivery of an Intervention to Promote Mental Health Among Latina Immigrant Women. J Integr Complement Med. 2022 Oct;28(10):821-829. doi: 10.1089/jicm.2022.0491. Epub 2022 Jun 20. PMID 35723668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two community-based organizations serving Latino immigrants over four waves between September 2018 - February 2021. Bilingual study team members and community organization staff recruited participants by promoting the study to clients via flyers, PowerPoint presentations, social media announcements and word of mouth.
Units Other Than Participants: Site
Groups:
- ALMA Intervention Group: Amigas Latinas Motivando el Alma (ALMA). This group receives the intervention after baseline assessment.
  Amigas Latinas Motivando el Alma (ALMA): In a series of 8 weekly sessions, the program uses a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. Over the course of the eight ALMA sessions, 25 women are (1) engaged in activities to identify coping strategies they are currently using and encouraged to continue to use them; (2) introduced to new coping strategies (e.g. mindfulness techniques, increased social ties and social support); and, (3) provided resources for seeking additional help if needed.
  Due to COVID-19 pandemic, the intervention was changed to online synchronous delivery via Zoom over 6 weekly sessions.
- ALMA Delayed Intervention Control Group: Amigas Latinas Motivando el Alma (ALMA). This group receives the intervention five months after the baseline assessment (after the post-intervention, and 3 month assessments have been completed).
  Amigas Latinas Motivando el Alma (ALMA): In a series of 8 weekly sessions, the program uses a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. Over the course of the eight ALMA sessions, 25 women are (1) engaged in activities to identify coping strategies they are currently using and encouraged to continue to use them; (2) introduced to new coping strategies (e.g. mindfulness techniques, increased social ties and social support); and, (3) provided resources for seeking additional help if needed.
  Due to COVID-19 pandemic, the intervention was changed to online synchronous delivery via Zoom over 6 weekly sessions.
Period: Overall Study
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
Started | 111; 1 Site | 115; 1 Site
Attended at Least One Session | 103; 1 Site | 85; 1 Site
Attended 50% of Sessions | 88; 1 Site | 65; 1 Site
Attended 75% of Intervention Sessions | 56; 1 Site | 57; 1 Site
Follow-up, 2 Months After Baseline | 99; 1 Site | 100; 1 Site
Follow-up, 4 Months After Baseline | 94; 1 Site | 103; 1 Site
Completed | 94; 1 Site | 103; 1 Site
Not Completed | 17; 0 Site | 12; 0 Site
Not completed — Lost to Follow-up | 15 | 10
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group | Total
Number analyzed (Participants) | 111 | 115 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 113 | 220
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.23 (1.04) | 39.09 (0.03) | 40.14 (0.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 115 | 226
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 115 | 226
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 96 | 89 | 185
  El Salvador | 6 | 5 | 11
  Colombia | 1 | 3 | 4
  Venezuela | 1 | 1 | 2
  Ecuador | 1 | 0 | 1
  Peru | 1 | 0 | 1
  Guatemala | 5 | 10 | 15
  Argentina | 0 | 1 | 1
  United States | 0 | 2 | 2
  Chile | 0 | 1 | 1
  Honduras | 0 | 2 | 2
  Bolivia | 0 | 1 | 1
Education, categorical [Count of Participants; unit: Participants]
  High school degree or higher | 67 | 83 | 150
  Less than high school degree | 44 | 32 | 76
Immigration status, categorical [Count of Participants; unit: Participants]
  Current visa/ permission | 24 | 37 | 61
  Entry and/or stay without permission | 73 | 59 | 132
  Preferred not to answer | 14 | 19 | 33
Anxiety symptoms, continuous [Mean (Standard Deviation); unit: units on a scale] — range of 0 (minimum) to 21 (maximum) with higher scores indicating more frequent symptoms of anxiety
  units on a scale | 6.67 (0.40) | 7.06 (0.40) | 6.87 (0.30)
Anxiety symptoms, categorical [Count of Participants; unit: Participants]
  None (0-4) | 39 | 37 | 76
  Mild (5-9) | 46 | 46 | 92
  Moderate (10-14) | 19 | 21 | 40
  Severe (15-21) | 7 | 11 | 18
Depressive symptoms, continuous [Mean (Standard Deviation); unit: units on a scale] — range of 0 (minimum) to 27 (maximum) with higher scores indicating more frequent symptoms of depression
  units on a scale | 7.06 (0.50) | 6.66 (0.40) | 6.86 (0.30)
Depressive symptoms, categorical [Count of Participants; unit: Participants]
  None (0-4) | 42 | 47 | 89
  Mild (5-9) | 41 | 39 | 80
  Moderate (10-14) | 15 | 20 | 35
  Moderate to Severe (15-27) | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Frequency of depressive symptoms as measured by the Patient Health Questionnaire 9 in the last two weeks. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Higher scores indicate a worse outcome.
Time Frame: Baseline, 2 months after baseline (post-intervention for intervention group), 4 months after baseline, and 6 months after baseline. Outcomes reported at baseline, 2 and 4 months after baseline for both intervention and control groups.
Population: In the intervention group: 12 participants were lost to follow-up at 2-month post-intervention time point, and 17 were not able to be contacted at the 4 month follow-up time point. In the control group: 15 participants were lost to follow-up at 2-month post intervention time point, and 12 were not able to be contacted at 4 month follow-up time point. Reasons were that they could not be contacted or declined to complete the survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
Number analyzed (Participants) | 111 | 115
score on a scale
  Baseline | 7.01 [6.10 to 7.92] | 6.61 [5.76 to 7.47]
  Two-month follow-up: number analyzed (Participants) | 99 | 100
  Two-month follow-up | 4.96 [4.06 to 5.87] | 6.39 [5.32 to 7.45]
  Four-month follow-up: number analyzed (Participants) | 94 | 103
  Four-month follow-up | 5.19 [4.20 to 6.18] | 6.31 [5.27 to 7.36]

2. Primary Outcome: Anxiety Symptoms
Description: Frequency of anxiety symptoms as measured by the General Anxiety Disorders 7 in the last two weeks. Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder (GAD). Scores range from 0 to 21. Scores ≥10. Anxiety Severity: 1-4 minimal symptoms, 5-9 mild symptoms, 10-14 moderate symptoms, 15-21 severe symptoms. Higher scores indicate a worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
Number analyzed (Participants) | 111 | 115
score on a scale
  Baseline | 6.71 [5.83 to 7.60] | 7.02 [6.17 to 7.86]
  Two-month follow-up: number analyzed (Participants) | 99 | 100
  Two-month follow-up | 4.09 [3.34 to 4.84] | 5.56 [4.67 to 6.46]
  Four-month follow-up: number analyzed (Participants) | 94 | 103
  Four-month follow-up | 4.30 [3.48 to 5.12] | 5.35 [4.43 to 6.27]

3. Secondary Outcome: Stress
Description: Frequency of perceived stress in the last month. The Perceived Stress Scale (PSS) is a classic stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. Higher scores indicate worse outcomes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
Number analyzed (Participants) | 111 | 115
score on a scale
  Baseline | 6.36 (0.30) | 6.27 (0.27)
  Two month follow-up: number analyzed (Participants) | 99 | 100
  Two month follow-up | 5.20 (0.25) | 5.65 (0.29)
  Four month follow-up: number analyzed (Participants) | 94 | 103
  Four month follow-up | 5.19 (0.33) | 5.73 (0.31)

4. Other Pre Specified Outcome: Program Satisfaction
Description: Survey items that ask participant about their level of satisfaction with the program. Response options of 1 - 5, with 5 indicating highest satisfaction (better outcome).
Time Frame: Assessed in the intervention group at post-intervention follow-up, 2 months after baseline. In the control group, it was assessed post-intervention, 6 months after baseline.
Population: In the intervention group: 14 participants were either lost to follow-up at two month time point or did not attend any sessions and therefore were not asked these questions. In the control group: 39 participants were either lost to follow-up at two month time point or did not attend any sessions and therefore were not asked the questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
Number analyzed (Participants) | 97 | 76
score on a scale
  Would recommend program | 4.95 (0.02) | 4.80 (0.05)
  Program was relevant | 4.84 (0.05) | 4.78 (0.05)
  Enjoyed ALMA program | 4.92 (0.03) | 4.71 (0.06)
  The program helped improve my mental health | 4.82 (0.04) | 4.63 (0.08)

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected through the final follow-up (9 months after baseline).
Description: Does not differ.
Arm/Group | ALMA Intervention Group | ALMA Delayed Intervention Control Group
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/115
Other Adverse Events (participants affected / at risk) | 0/111 | 0/115

LIMITATIONS AND CAVEATS:
Half of trial had to be conducted under COVID-19 protocol which changed intervention delivery and modes of data collection (phone instead of in-person).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03545282/Prot_SAP_000.pdf